CLINICAL TRIAL: NCT06362343
Title: The Study of Monitoring and Dosing Guidance of Direct Oral Anticoagulants Based on Pharmacokinetics, Pharmacodynamics, and Pharmacogenomics
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Ruijin Hospital (Other); Xiangya Hospital of Central South University (Other); China-Japan Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-Rivaroxaban-Monitoring
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood（Cells and Plasma）and Urine
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with pulmonary embolism and using direct oral anticoagulants: Patients with pulmonary embolism and using direct oral anticoagulants
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban

SUMMARY:
1. Integrate pharmacokinetic-pharmacodynamic (PK-PD) modeling and pharmacogenomics techniques to develop a population PK-PD model, aiming to explore monitoring and dose guidance schemes for Direct Oral Anticoagulants (DOACs).
2. Investigate the factors influencing PK-PD of DOACs in the pulmonary embolism population, clarifying the correlation between genotype characteristics and clinical outcomes.
3. Explore the correlation between drug concentrations, coagulation indices, and clinical outcomes of DOACs, defining the indications for DOACs testing and the overall monitoring process.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with acute symptomatic pulmonary embolism objectively diagnosed by imaging (with or without deep vein thrombosis) who have completed anticoagulation for the acute phase and have entered the maintenance phase of anticoagulation
* Expected lifespan greater than 3 months
* Eligible for the use of Xa factor inhibitors;
* Agreement to participate in the study, signing of informed consent, and commitment to regular follow-up.

Exclusion Criteria:

* Moderate or severe liver dysfunction (Child-Pugh grade B or C);
* Severe renal impairment (CrCl < 15 ml/min);
* Pregnant or breastfeeding women;
* Tendency for spontaneous bleeding, such as coagulopathy or thrombocytopenia (PLT < 20×10^9/L);
* Contraindications for the use of other Xa factor inhibitors;
* Patients diagnosed with hereditary thrombophilia and antiphospholipid syndrome.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pulmonary embolism and are using DOACs.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Bleeding events | Through the entire follow-up time, 3 months
  Major bleeding events, clinical relatied non-major bleeding events and minor bleeding events
Recurrent thromboembolic events | Through the entire follow-up time, 3 months
  Recurrent thromboembolic events

CONTACTS AND LOCATIONS:
Overall Officials: Juhong Shi, M.D, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
If there is a reasonable data request, you can contact the project leader via email to obtain the data.